CLINICAL TRIAL: NCT01885949
Title: Phase 2 Combination Trial of Tivozanib and Enzalutamide in Men With Advanced Prostate Cancer
Brief Title: Tivozanib + Enzalutamide in Adv Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Dror Michaelson, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-073
Record Dates: First submitted 2013-06-19; First posted 2013-06-25 (Estimated); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Metastatic
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — tivozanib; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Treatment Arm (Experimental): Tivozanib, taken daily for 21 days followed by a 7 day break Enzalutamide taken daily for 28 days
  Interventions: Drug: Tivozanib; Drug: Enzalutamide

INTERVENTIONS:
Drug: Tivozanib — Oral
  Other Names: AV-951
Drug: Enzalutamide — oral
  Other Names: MDV-3100

SUMMARY:
This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational combination of drugs to learn whether they work in treating a specific cancer. "Investigational" means that the combination of drugs is still being studied and that research doctors are trying to find out more about it, such as the safest dose to use and the side effects they may cause. It also means that the FDA has not yet approved the combination.

The two drugs being tested in this study are tivozanib and enzalutamide. Enzalutamide has been approved by the FDA for treatment of prostate cancer. On the other hand, tivozanib is still investigational, and has not been tested in a combination with enzalutamide before.

Enzalutamide is an androgen receptor antagonist (it blocks the activity of the male sex hormones). Prostate cancers are initially dependent on the male hormone testosterone for growth. Hormonal therapies that lower testosterone or block the ability of testosterone to act at the level of the prostate cancer are currently among the most effective treatments for prostate cancers taht have spread to other body organs (metastasized). The effectiveness of hormonal treatments, however, is not permanent, and over time many prostate cancers progress in spite of these treatments. Enzalutamide is a drug that has been proven to help delay the progression of advanced prostate cancer on average for about 8 months.

Tivozanib is an anti-angiogenesis medicine that fights different types of cancer by blocking the blood supply to the tumor, so that the tumor does not receive the nutrients it needs to grow. The main goal of this study is to determine whether the combination of tivozanib and enzalutamide is more effective in delaying the progression of disease than when enzalutamide is given alone. This study will also determine whether treatment with the combination of the tivozanib and enzalutamide will have more side effects then treatment with enzalutamide alone.

DETAILED DESCRIPTION:
Patients will be treated in treatment cycles of 28 days (4 weeks), during which time they will take tivozanib once a day for 21 days (3 weeks) followed by a one week break from treatment. The other medication, enzalutamide, will be taken every day throughout each cycle.

Patients will be given a Study Drug Administration Diary to keep a brief record of medication administration, and to record any side effects or symptoms.

Patients will be seen in the clinic at the beginning of each cycle (every 4 weeks). During each visit they will have the following procedures: medical history, vital sign measurements, complete physical examination, performance status, routine blood tests, urine sample, prostate specific antigen (PSA) test, assessment of tumor, review of study drug administration diary, and review of current medications.

About four weeks after stopping the study drug patients will be asked to return to the research clinic for a final study visit. The following procedures will be done: medical history, vital sign measurements, brief physical examination, electrocardiogram, review of other medications used since the last visit, routine blood tests, urine sample and a review of any changes in health.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate that is metastatic or unresectable and for which standard curative options do not exist
* Radiographic evidence of metastatic prostate cancer
* Progressive disease despite ongoing androgen deprivation therapy (ADT), defined as castration resistant prostate cancer (CRPC)
* Other than ongoing prior treatment with other hormonal agents such as antiandrogens or ketoconazole must have been stopped at least two weeks prior to enrollment
* Have received prior docetaxel-based chemotherapy for prostate cancer within the past 12 months. Such chemotherapy must have been stopped at least 3 weeks prior to the first dosing in this study
* Life expectancy of at least 12 weeks
* Must agree to use adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

* Prior treatment with enzalutamide, TOK-001, or ARN-509
* Participants who have received more than two prior chemotherapy regimens for metastatic CRPC
* Receiving any other investigational anticancer agents
* Known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tivozanib or enzalutamide
* Radiotherapy or minor surgical procedure within 2 weeks, or major surgical procedure within 4 weeks prior to administration of first dose of study drug; inadequate recovery from prior surgical procedure
* History of seizure of condition that may predispose to seizure
* Significant cardiovascular disease
* Non-healing wound, bone fracture or skin ulcer
* Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis or other gastrointestinal condition with increased risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to administration of first dose of study drug
* Serious/active infection or infection requiring parenteral antibiotics
* Significant thromboembolic or vascular disorders within 6 months prior to administration of first dose of study drug
* Currently active second primary malignancy, including hematologic malignancies, except for non-melanoma skin cancers, in situ cervical cancer, and ductal or lobular carcinoma in situ of the breast
* History of genetic or acquired immune suppression disease such as HIV; subjects on immune suppressive therapy for organ transplant
* Inability to swallow capsules, malabsorption syndrome or gastrointestinal disease that severly affects the absorption of study drugs, major resection of the stomach or small bowel, or gastric bypass procedure
* Significant bleeding disorders within 6 months prior to administration of first dose of study drug
* Psychiatric disorder or altered mental status precluding informed consent or protocol-related testing

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-09-03 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Dror Michaelson, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Treatment Arm
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Treatment Arm
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: The primary objective of this study will be to demonstrate an improvement in progression free survival in men with metastatic castration resistant prostate cancer (mCRPC) treated with tivozanib and enzalutamide.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Experimental Treatment Arm
Number analyzed (Participants) | 5
participants | 5

2. Secondary Outcome: Safety and Tolerability
Description: Safety and tolerability of tivozanib and enzalutamide will be assessed. The number of patients having grades 1-4 adverse events by NCI CTC version 4.0 will be recorded.
Time Frame: 2 years
Population: No Grade 3/4 SAEs
Measure: Number; unit: events
Arm/Group | Experimental Treatment Arm
Number analyzed (Participants) | 5
events | 0

3. Secondary Outcome: Overall Survival
Description: To estimate overall survival in patients treated with tivozanib and enzalutamide
Time Frame: 2 years
Population: Insufficient patients enrolled to allow statistical analysis of overall survival
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Arm
Number analyzed (Participants) | 5
Participants | 5

4. Secondary Outcome: PSA Response Rate
Description: To evaluate PSA response rate
Time Frame: 2 years
Population: Insufficient number of patients to allow statistical analysis of data
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Arm
Number analyzed (Participants) | 5
Participants | 5

5. Secondary Outcome: Time to PSA Progression
Description: The time to PSA progression (in months) will be evaluated in patients treated with enzalutamide and tivozanib
Time Frame: 2 years
Population: Insufficient number of patients to allow statistical analysis of data
Measure: Median (Standard Deviation); unit: months
Arm/Group | Experimental Treatment Arm
Number analyzed (Participants) | 5
months | 12 (6)

ADVERSE EVENTS:
Time Frame: 2 years
Description: No grade 3/4 SAEs reported
Arm/Group | Experimental Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT01885949/Prot_SAP_000.pdf